CLINICAL TRIAL: NCT04328454
Title: Clinical Characteristics and Prognostic Factors of Patients With COVID-19 in Chibi Hospital of Hubei Province
Brief Title: Clinical Characteristics and Prognostic Factors of Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Chibi People's Hospital, Hubei Province (Unknown)
Responsible Party: Principal Investigator, Ming Li, Shanghai 10th People's Hospital, Shanghai 10th People's Hospital
Other Study IDs: HBCBH-IEC-2020-101
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: Hospitalized patients with COVID-19
  Interventions: Other: retrospective analysis

INTERVENTIONS:
Other: retrospective analysis — The investigators retrospectively analyzed the hospitalized patients with COVID-19

SUMMARY:
As of February 17th, 2020, China has 70635 confirmed cases of coronavirus disease 2019 (COVID-19), including 1772 deaths. Human-to-human spread of virus via respiratory droplets is currently considered to be the main route of transmission. The number of patients increased rapidly but the impact factors of clinical outcomes among hospitalized patients are still unclear.

DETAILED DESCRIPTION:
As of February 17th, 2020, China has 70635 confirmed cases of coronavirus disease 2019 (COVID-19), including 1772 deaths. Human-to-human spread of virus via respiratory droplets is currently considered to be the main route of transmission. The number of patients increased rapidly but the impact factors of clinical outcomes among hospitalized patients are still unclear.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged >=18years old; Diagnosed with CONVID19. Diagnostic criteria including: Laboratory (RT-PCR) confirmed SARS-Cov-2 infection; CT of the lung conformed to the manifestation of viral pneumonia.

Exclusion Criteria:

* Near-death state (expected survival time less than 24 hours); Malignant tumor; Pregnancy or puerperium women; Patients who refused to participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-04-02 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
Time to negative conversion of severe acute respiratory syndrome coronavirus 2 | 1 month
  The primary outcome is the time to negative conversion of coronavirus

SECONDARY OUTCOMES:
Length of stay in hospital | 1 month
  The time of hospitalization
Survival | 1 month
  The rate of survival within hospitalization of these patients will be tracked. The rate of survival within hospitalization of these patients will be tracked. The rate of survival within hospitalization of these patients will be tracked. The rate of survival within hospitalization of these patients will be tracked.
Intubation | 1 month
  The rate of intubation within hospitalization of these patients will be tracked

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No